CLINICAL TRIAL: NCT03028363
Title: A Randomized, Double-blind, Vehicle Controlled, Efficacy and Safety Study of Olumacostat Glasaretil Gel in Subjects With Acne Vulgaris
Brief Title: A Study of Olumacostat Glasaretil Gel in Subjects With Acne Vulgaris
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dermira, Inc. (Industry)
Responsible Party: Sponsor
Organization: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DRM01B-ACN03
Record Dates: First submitted 2017-01-19; First posted 2017-01-23 (Estimated); Results first posted 2019-02-05 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Olumacostat Glasaretil Gel, 5.0% (Experimental): Olumacostat Glasaretil Gel, 5.0%, applied twice daily to the face for 12 weeks
  Interventions: Drug: Olumacostat Glasaretil Gel, 5.0%
- Olumacostat Glasaretil Gel, Vehicle (Placebo Comparator): Olumacostat Glasaretil Gel, Vehicle, applied twice daily to the face for 12 weeks
  Interventions: Other: Olumacostat Glasaretil Gel, Vehicle

INTERVENTIONS:
Drug: Olumacostat Glasaretil Gel, 5.0% — Gel containing Olumacostat Glasaretil
  Other Names: DRM01
  Arms: Olumacostat Glasaretil Gel, 5.0%
Other: Olumacostat Glasaretil Gel, Vehicle — Vehicle (placebo) gel
  Arms: Olumacostat Glasaretil Gel, Vehicle

SUMMARY:
The objectives of this study are to assess the safety and efficacy of Olumacostat Glasaretil Gel compared to vehicle in patients with acne vulgaris

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent and, for subjects under legal adult age, signed assent
* Age ≥ 9 years
* Clinical diagnosis of facial acne vulgaris defined as:

  * At least 20 inflammatory lesions, and
  * At least 20 non-inflammatory lesions, and
  * Investigator Global Assessment of 3 or greater

Exclusion Criteria:

* Active cystic acne or acne conglobata, acne fulminans, and secondary acne
* Two or more active nodulocystic lesions on the face
* Clinically significant abnormal laboratory or ECG result
* Subjects who are actively participating in an experimental therapy study or who have received experimental therapy within 30 days or 5 half-lives (whichever is longer) of the Baseline visit
* Treatment with over-the-counter topical medications for the treatment of acne vulgaris including benzoyl peroxide, topical anti-inflammatory medications, corticosteroids, α-hydroxy/glycolic acid on the face within 2 weeks prior to Baseline
* Treatment with systemic antibiotics or systemic anti-acne drugs or topical retinoid within 4 weeks prior to Baseline
* Treatment with a new hormonal therapy or dose change to existing hormonal therapy within 12 weeks prior to Baseline (hormonal therapies include, but are not limited to, estrogenic and progestational agents such as birth control pills).
* Use of androgen receptor blockers (such as spironolactone or flutamide) within 2 weeks prior to Baseline.
* Oral retinoid use (e.g., isotretinoin) within 12 months prior to Baseline or vitamin A supplements greater than 10,000 units/day within 6 months prior to Baseline
* Facial procedures (chemical or laser peel, microdermabrasion, etc.) within the past 8 weeks

Min Age: 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 759 (Actual)
Dates: Start 2016-12-27 (Actual); Primary Completion 2017-11-28 (Actual); Study Completion 2017-11-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Beth Zib, Study Director — Dermira, Inc.
Locations (49):
- United States (38):
  - Alliance Dermatology & MOHS Center, Phoenix, Arizona
  - Anaheim Clinical Trials, Anaheim, California
  - Dermatology Research Associates, Los Angeles, California
  - Rady Children's Hospital UCSD Pediatric and Adolescent Derm, San Diego, California
  - University Clinical Trials Inc., San Diego, California
  - Horizons Clinical Research Center, LLC, Denver, Colorado
  - Dermatology Physicians of CT, Shelton, Connecticut
  - Finlay Medical Research, Miami, Florida
  - Health Awareness, Inc, Port Saint Lucie, Florida
  - International Clinical Research-US, LLC, Sanford, Florida
  - Lenus Research & Medical Group, Sweetwater, Florida
  - Research Institute of the Southeast, LLC, West Palm Beach, Florida
  - Arlington Dermatology, Arlington Heights, Illinois
  - Forefront Dermatology, Carmel, Indiana
  - Kansas City Dermatology, PA, Overland Park, Kansas
  - Skin Sciences, PLLC, Louisville, Kentucky
  - Lawrence Jeffrey Green MD, LLC, Rockville, Maryland
  - Great Lakes Research Group, Inc, Bay City, Michigan
  - Minnesota Clinical Study Center, Fridley, Minnesota
  - Mercy Research, Washington, Missouri
  - Meridian Clinical Research, LLC, Norfolk, Nebraska
  - Quality Clinical Research Inc, Omaha, Nebraska
  - Meridian Clinical Research, Omaha, Nebraska
  - Acne Treatment & Research Center, Morristown, New Jersey
  - Schweiger Dermatology, PLLC, New York, New York
  - DermResearchCenter of New York, Inc., Stony Brook, New York
  - Cyn3rgy Research, Gresham, Oregon
  - Clinical Partners, LLC, Johnston, Rhode Island
  - Meridian Clincial Research, Dakota Dunes, South Dakota
  - International Clinical Research - Tennessee LLC, Murfreesboro, Tennessee
  - International Clinical Research-Tennesse LLC, Murfreesboro, Tennessee
  - DermResearch, Austin, Texas
  - J &S Studies, Inc, College Station, Texas
  - Synexus US, LP, dba, Research Across America, Murphy, Texas
  - Progressive Clinical Research, PA, San Antonio, Texas
  - Clinical Trials of Texas, Inc., San Antonio, Texas
  - Dermatology Clinical Research Center of San Antonio, San Antonio, Texas
  - Virginia Clinical Research, Inc., Norfolk, Virginia
- Australia (5):
  - Woden Dermatology, Phillip, Australian Capital Territory
  - St George Dermatology and Skin Cancer Centre, Kogarah, New South Wales
  - North Eastern Health Specialists, Hectorville, South Australia
  - Skin & Cancer Foundation Inc., Carlton, Victoria
  - Fremantle Dermatology, Fremantle, Western Australia
- Canada (6):
  - Institute for Skin Advancement, Calgary, Alberta
  - SimcoDerm Medical and Surgical Dermatology Center, Barrie, Ontario
  - Lynderm Research Inc., Markham, Ontario
  - North Bay Dermatology Centre, North Bay, Ontario
  - Research Toronto, Toronto, Ontario
  - Windsor Research Inc., Windsor, Ontario

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Olumacostat Glasaretil Gel, 5.0% | Olumacostat Glasaretil Gel, Vehicle
Started | 498 | 261
Completed | 420 | 228
Not Completed | 78 | 33

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Olumacostat Glasaretil Gel, 5.0% | Olumacostat Glasaretil Gel, Vehicle | Total
Number analyzed (Participants) | 498 | 261 | 759
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 289 | 140 | 429
  Between 18 and 65 years | 209 | 121 | 330
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 19.4 (6.58) | 20.1 (7.14) | 19.7 (6.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 286 | 152 | 438
  Male | 212 | 109 | 321
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 150 | 68 | 218
  Not Hispanic or Latino | 346 | 193 | 539
  Unknown or Not Reported | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 3 | 6
  Asian | 13 | 11 | 24
  Native Hawaiian or Other Pacific Islander | 3 | 0 | 3
  Black or African American | 79 | 43 | 122
  White | 373 | 191 | 564
  More than one race | 27 | 13 | 40
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 32 | 16 | 48
  United States | 431 | 226 | 657
  Australia | 35 | 19 | 54
Fitzpatrick Skin Type [Count of Participants; unit: Participants] — Fitzpatrick Skin Type is a scale to numerically classify skin color, defined by the response to ultraviolet (UV) light with the following categories:
  Type I Burns easily, rarely tans Type II Burns easily, tans minimally Type III Burns moderately, tans gradually Type IV Burns minimally, tans well Type V Rarely burns, tans profusely Type VI Never burns, deeply pigmented
  Participants
    Type I | 28 | 16 | 44
    Type II | 94 | 55 | 149
    Type III | 125 | 75 | 200
    Type IV | 115 | 55 | 170
    Type V | 79 | 29 | 108
    Type VI | 57 | 31 | 88

OUTCOME MEASURES:

1. Primary Outcome: Mean Absolute Change in Acne Lesion Counts (Inflammatory) From Baseline to Week 12
Description: Mean absolute change in acne lesion counts (inflammatory) from baseline to Week 12
Time Frame: Baseline and Week 12
Population: Intent-to-Treat
Measure: Least Squares Mean (Standard Deviation); unit: Lesions
Arm/Group | Olumacostat Glasaretil Gel, 5.0% | Olumacostat Glasaretil Gel, Vehicle
Number analyzed (Participants) | 498 | 261
Lesions | -14.5 (14.85) | -13.5 (14.54)
Statistical Analysis 1: Comparison: Olumacostat Glasaretil Gel, 5.0% vs Olumacostat Glasaretil Gel, Vehicle; Test type: Other; p = 0.3430, ANCOVA; Ranked ANCOVA, Markov Chain Monte Carlo (MCMC) Multiple Imputation

2. Primary Outcome: Mean Absolute Change in Acne Lesion Counts (Non-inflammatory) From Baseline to Week 12
Description: Mean absolute change in acne lesion counts (non-inflammatory) from baseline to Week 12
Time Frame: Baseline and Week 12
Population: Intent-to-Treat
Measure: Least Squares Mean (Standard Deviation); unit: Lesions
Arm/Group | Olumacostat Glasaretil Gel, 5.0% | Olumacostat Glasaretil Gel, Vehicle
Number analyzed (Participants) | 498 | 261
Lesions | -14.1 (21.05) | -11.8 (20.28)
Statistical Analysis 1: Comparison: Olumacostat Glasaretil Gel, 5.0% vs Olumacostat Glasaretil Gel, Vehicle; Test type: Other; p = 0.1260, ANCOVA; Ranked ANCOVA, Markov Chain Monte Carlo (MCMC) Multiple Imputation

3. Primary Outcome: Percentage of Subjects Who Achieved ≥ 2-grade Improvement and a Grade of 0 or 1 in the Investigator Global Assessment of Acne (IGA) From Baseline to Week 12
Description: Percentage of subjects who achieved ≥ 2-grade improvement and a grade of 0 or 1 in the investigator global assessment of acne (IGA) from baseline to Week 12
  Scoring Criteria for Investigator Global Assessment 0 - Clear skin with no inflammatory or noninflammatory lesions
  1. - Almost clear; rare noninflammatory lesions with no more than one small inflammatory lesion
  2. - Mild severity; greater than Grade 1; some noninflammatory lesions with no more than a few inflammatory lesions (papules/pustules only, no nodular lesions)
  3. - Moderate severity; greater than Grade 2; up to many noninflammatory lesions and may have some inflammatory lesions, but no more than one small nodular lesion
  4. - Severe; greater than Grade 3; up to many noninflammatory and inflammatory lesions, but no more than a few nodular lesions
Time Frame: Baseline and Week 12
Population: Intent-to-Treat
Measure: Count of Participants; unit: Participants
Arm/Group | Olumacostat Glasaretil Gel, 5.0% | Olumacostat Glasaretil Gel, Vehicle
Number analyzed (Participants) | 498 | 261
Participants
  Success | 95 | 54
  Failure | 403 | 207
Statistical Analysis 1: Comparison: Olumacostat Glasaretil Gel, 5.0% vs Olumacostat Glasaretil Gel, Vehicle; Test type: Other; p = 0.5247, Regression, Logistic; Logistic Regression (Firth's Penalized Likelihood), MCMC Multiple Imputation

ADVERSE EVENTS:
Time Frame: Baseline to Week 12
Description: The Total Participants at risk are based on the Safety Population defined as Participants who were randomized and received at least one confirmed dose of study drug.
Arm/Group | Olumacostat Glasaretil Gel, 5.0% | Olumacostat Glasaretil Gel, Vehicle
All-Cause Mortality (participants affected / at risk) | 0/485 | 0/258
Serious Adverse Events (participants affected / at risk) | 1/485 | 3/258
Other Adverse Events (participants affected / at risk) | 89/485 | 33/258
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Olumacostat Glasaretil Gel, 5.0% (N=485) | Olumacostat Glasaretil Gel, Vehicle (N=258)
Constipation (Gastrointestinal disorders) | 0 | 1
Appendicitis (Infections and infestations) | 0 | 1
Epilepsy (Nervous system disorders) | 1 | 0
Bipolar disorder (Psychiatric disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Olumacostat Glasaretil Gel, 5.0% (N=485) | Olumacostat Glasaretil Gel, Vehicle (N=258)
Application site dryness (General disorders) | 13 | 2
Application site erythema (General disorders) | 13 | 3
Application site pain (General disorders) | 19 | 11
Application site pruritus (General disorders) | 13 | 4
Nasopharyngitis (Infections and infestations) | 15 | 5
Upper respiratory tract infection (Infections and infestations) | 16 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2016-10-06): https://cdn.clinicaltrials.gov/large-docs/63/NCT03028363/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-19): https://cdn.clinicaltrials.gov/large-docs/63/NCT03028363/SAP_001.pdf